CLINICAL TRIAL: NCT03004781
Title: Stimulation of Parents' Self-efficacy Beliefs and Emotion Coaching Practices to Reduce Externalizing Behavior in Preschoolers
Brief Title: Stimulation of Parents' Self-efficacy Beliefs and Emotion Coaching Practices (H2M1)
Acronym: H2M1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Isabelle Roskam, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLouvain_H2M1
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Behavior Problem
Keywords: parenting intervention; externalizing behavior; emotion coaching practices; self-efficacy beliefs
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Waiting-list (No Intervention): 8-week period without intervention, N=45
- self-efficacy (Experimental): 8-week group-based parenting program on self-efficacy beliefs, N=19
  Interventions: Behavioral: Parenting program
- self-efficacy/emotion coaching (Experimental): 8-week group-based parenting program on self-efficacy beliefs and emotion coaching practice, N=26
  Interventions: Behavioral: Parenting program

INTERVENTIONS:
Behavioral: Parenting program
  Arms: self-efficacy; self-efficacy/emotion coaching

SUMMARY:
This research compared the efficacy of two parenting interventions that vary according to the number and the nature of variables in reducing preschoolers' externalizing behavior (EB). The goal was to identify which parenting intervention format (one-variable versus two-variable) caused higher behavioral adjustment in children.

DETAILED DESCRIPTION:
The first format was a one-variable intervention manipulating parental self-efficacy beliefs. The second format was a two-variable intervention manipulating both parents' self-efficacy beliefs and emotion coaching practices. The two interventions shared exactly the same design, consisting of eight parent group sessions. Effect on children's EB and observed behaviors were evaluated through a multi-method assessment at three points (pre-test, post-test and follow-up).

ELIGIBILITY:
Inclusion Criteria:

* children in the clinical or borderline range of the EB scale (cut-off = 21 or higher) of the Child Behavior Checklist preschool form (Achenbach & Rescorla, 2000a)
* three to six years old and still in kindergarten at the beginning of the intervention

Exclusion Criteria:

* children with intellectual disabilities (average IQ < 5.5)
* highly gifted children (average IQ >14.5)

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in child behavior | 0 week, 8 weeks, 24 weeks
  parent reports of child behavior and standardized observation of parent-child interaction

SECONDARY OUTCOMES:
Change in parental self-efficacy beliefs | 0 week, 8 weeks, 24 weeks
  parent questionnaire
Change in parenting behavior | 0 week, 8 weeks, 24 weeks
  standardized observation of parent-child interaction

IPD SHARING:
Plan to Share IPD: No